CLINICAL TRIAL: NCT05289323
Title: Evaluation of Intrathecal Neostigmine as an Adjuvant to Bupivacaine in Ameliorating Post-Dural Puncture Headache in Elective Caesarian Section: A Prospective Randomized Controlled Clinical Trial
Brief Title: Effect of Intrathecal Neostigmine on Post-dural Puncture Headache.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Kasr El Aini Hospital (Other); Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Elnaggar, Principal Investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB NO: 00012098 SN: 0305408
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Post-Dural Puncture Headache
Keywords: Neostigmine; Intrathecal; prevention of PDPH; PDPH; Caesarean section
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Neostigmine; Glucose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Intervention group (N) (Experimental): 0.5 mg ampule (1 ml) will be diluted in 4 ml dextrose 5% to make a solution of 100 μg/ml, 0.2 ml of this solution will be added to 2.5 ml of hyperbaric bupivacaine 0.5 % used for intrathecal injection.
  Interventions: Drug: Neostigmine Methylsulfate
- The control group (C) (Placebo Comparator): one ml of normal saline 0.9 % will be mixed with 4 ml dextrose 5 % in the five-milliliter syringe. 0.2 ml of this mixture will be added to 2.5 ml of hyperbaric bupivacaine 0.5 % used for intrathecal injection.
  Interventions: Drug: Dextrose 5%/Nacl 0.9% Inj

INTERVENTIONS:
Drug: Neostigmine Methylsulfate — 0.5 mg ampule (1 ml) will be diluted in 4 ml dextrose 5% to make a solution of 100 μg/ml, 0.2 ml of this solution will be added to 2.5 ml of hyperbaric bupivacaine 0.5 % used for intrathecal injection.
  Other Names: Neostigmine 20 mic
  Arms: The Intervention group (N)
Drug: Dextrose 5%/Nacl 0.9% Inj — one ml of normal saline 0.9 % will be mixed with 4 ml dextrose 5 % in the five-milliliter syringe. 0.2 ml of this mixture will be prepared at a one-milliliter identical syringe.
  Other Names: Dextrose 5 %Nacl0.9%
  Arms: The control group (C)

SUMMARY:
Intravenous neostigmine was recently reported as an effective treatment for PDPH for parturients after intrathecal (IT) block which is postulated to be through its central effects on CSF secretion and cerebral vascular tone modulation. Intrathecal neostigmine has been investigated widely and found to be an effective adjuvant to bupivacaine for postoperative analgesia.

The objective of the current study is to investigate the possible prophylactic role of intrathecal neostigmine as an adjuvant to bupivacaine in reducing the incidence and severity of post-dural puncture headache in parturients scheduled for an elective cesarean section.

DETAILED DESCRIPTION:
Upon arrival to the operating room standard monitors will be applied and continued all over the operation, an 18G peripheral intravenous (IV) cannula will be inserted, and 15 ml/kg of Ringer lactate solution will be infused.

The intrathecal block will be performed via a midline approach into the L3-4 or L4-5 interspaces in a sitting position under strict aseptic condition using a 25-gauge spinal needle after administration of 3 ml of lidocaine 2% (60 mg) as a subcutaneous infiltration, a 2.5 ml of hyperbaric bupivacaine, 0.5 % (12.5 mg) in addition to the content of the prepared study syringe will be mixed and slowly injected.

After ensuring sufficient anesthesia level by loss of sensation to pinprick at the T4 level, the surgical procedure will start with continuous hemodynamic monitoring and recording.

At the end of the surgery, the parturient will be transferred to the postoperative anesthesia care unit (PACU).

Parturients will be transferred to the obstetrics ward after fulfilling the criteria of the modified Aldrete scoring system ≥9.

The participants who will be diagnosed to have PDPH Per the previously mentioned criteria will be treated by using oral Panadol extra™ (paracetamol 1gm + caffeine 135 mg) (Manufactured by: Alexandria company for pharmaceuticals & chemical industries under license: GlaxoSmithKline Consumer Healthcare Ltd. Ireland) at 6-hour interval in addition to ensuring good oral or intravenous hydration (2-3 L/day) and bed rest. Severe Intractable headache (VAS ≥ 4) persistent for more than 48 hours with no response to conservative measures will be managed with an autologous epidural blood patch after participant approval and consent signing.

Assessment of the quality of the sensory and motor block in terms of the onset and duration will be done at 2 minutes intervals during the first 10 minutes after giving the spinal block, then at 10 minutes intervals until the end of the surgery, and at 15 minutes intervals while being in the PACU.

ELIGIBILITY:
Inclusion Criteria:

* American society association (ASA) physical status class II parturients with a single fetus who will be scheduled for an elective caesarian section by Intrathecal block.

Exclusion Criteria:

* Body mass index more than or equal to 35 kg/m2.
* Any contraindication to Intrathecal blocks such as local infection, bleeding disorders, or parturient refusal.
* Allergy to neostigmine or other drugs will be used in the study.
* Long-term opioid use.
* A history of chronic pain, migraine, cluster headache.
* Digestive problems with nausea and vomiting; cognitive dysfunction or memory disorders.
* Significant renal, hepatic, and cardiovascular diseases.
* History of urinary retention or bronchial asthma.
* Inadequate or failed Intrathecal block.
* Complicated pregnancy such as hypertensive disorders of the pregnancy, abnormal placenta, or uterine atony.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 722 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of post-dural puncture headache | Two times daily for five days after intrathecal block.
  any headache that develops within five days of dural puncture and can't be attributed to any other types of headache and mostly is postural in character.usually associated with neck stiffness, nausea, photophobia, and subjective hearing symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Gamal Eldine, MD, Study Director — University of Alexandria; Ahmed I Elnaggar, MD, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Result] Arevalo-Rodriguez I, Ciapponi A, Munoz L, Roque i Figuls M, Bonfill Cosp X. Posture and fluids for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2013 Jul 12;(7):CD009199. doi: 10.1002/14651858.CD009199.pub2. PMID 23846960
- [Result] Grant R, Condon B, Hart I, Teasdale GM. Changes in intracranial CSF volume after lumbar puncture and their relationship to post-LP headache. J Neurol Neurosurg Psychiatry. 1991 May;54(5):440-2. doi: 10.1136/jnnp.54.5.440. PMID 1865208
- [Result] Abdelaal Ahmed Mahmoud A, Mansour AZ, Yassin HM, Hussein HA, Kamal AM, Elayashy M, Elemady MF, Elkady HW, Mahmoud HE, Cusack B, Hosny H, Abdelhaq M. Addition of Neostigmine and Atropine to Conventional Management of Postdural Puncture Headache: A Randomized Controlled Trial. Anesth Analg. 2018 Dec;127(6):1434-1439. doi: 10.1213/ANE.0000000000003734. PMID 30169405
- [Result] Prabhakar A, Lambert T, Kaye RJ, Gaignard SM, Ragusa J, Wheat S, Moll V, Cornett EM, Urman RD, Kaye AD. Adjuvants in clinical regional anesthesia practice: A comprehensive review. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):415-423. doi: 10.1016/j.bpa.2019.06.001. Epub 2019 Jul 2. PMID 31791560
- [Result] Aldrete JA. Modifications to the postanesthesia score for use in ambulatory surgery. J Perianesth Nurs. 1998 Jun;13(3):148-55. doi: 10.1016/s1089-9472(98)80044-0. PMID 9801540
- [Result] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Result] Cesarini M, Torrielli R, Lahaye F, Mene JM, Cabiro C. Sprotte needle for intrathecal anaesthesia for caesarean section: incidence of postdural puncture headache. Anaesthesia. 1990 Aug;45(8):656-8. doi: 10.1111/j.1365-2044.1990.tb14392.x. PMID 2400077
- [Result] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823